CLINICAL TRIAL: NCT05263440
Title: A Pilot Study of the Immediate Effects of DLPFC tDCS on Attention Bias in Depression
Brief Title: Immediate Effects of DLPFC tDCS on Attention Bias
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started because one of the collaborators was not able to attend to the study requirements.
Sponsor: Johns Hopkins University (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00312231
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Female participants with Depression (Experimental): Female participants with mild to severe depression to determine if a single-session of tDCS can alter negative attention bias. The primary objective is to study if single-session tDCS will affect attention bias in depression and is not meant to treat depression.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Participants will complete a single 30 minutes tDCS session targeting the left DLPFC while sitting in a comfortable position. At the end of the tDCS session possible side effects experienced during the tDCS session will be recorded along with their intensity (rated using the visual analogue scale, 0-10) and duration. The session can be aborted at any time for any reason if the participant wishes.The MINDD STIM tDCS system is composed of a management component, treatment module, single-use sponge patches and supporting patches, a headband to hold in position the sponge patches, and 2 cables. A trained study technician will program the stimulation device through the management component setting to the following stimulation parameters:Stimulation intensity: 2.0 mA or 1.5 mA; Stimulation duration: 30 minutes;Ramp up duration: 30 seconds (beginning of stimulation);Ramp down duration: 30 seconds (end of stimulation)

SUMMARY:
This research is being done to test if the investigators can modify or reduce negative attention bias in depression following a single session of transcranial direct current stimulation (tDCS) over the left anodal dorsolateral prefrontal cortex (DLPFC) in patients with mild to severe depression. The study will consist of a single-session tDCS session administered onsite at the Johns Hopkins University (JHU). After the consent process, participants will complete the study (approximately one hour in duration) with the guidance of a research associate.

DETAILED DESCRIPTION:
This prospective pilot study will recruit 25 female participants, ages 18-45 (inclusive), with mild to severe depression (based on BDI-II score range 14-19 for mild and 29-63 for severe) to determine if a single-session of tDCS can alter negative attention bias. The primary objective is to study if single-session tDCS will affect attention bias in depression and is not meant to treat depression. Subjects may or may not be receiving treatment for mild-severe depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* Female
* Mild to severe depression (determined by BDI-II scores of 14-19 and 29-63, respectively)
* If taking antidepressants, medication must be stable ≥ 30 days prior to screening

Exclusion Criteria:

* Wide-Range Achievement Test-Fourth Edition (WRAT-4) Reading Subtest standard score <85 (to ensure understanding of test procedures)
* Insufficient visual and motor ability to operate the intervention and assessments as judged by treating neurologist or study staff
* Primary psychiatric disorder other than depression (based on MINI)
* Primary neurologic condition that would prevent ability to participate (as determined by study clinician).
* History of head trauma in the last year
* Medical device implants in the head or neck
* History or current uncontrolled seizure disorder
* Current substance abuse disorder
* Pregnant or lactating women
* Skin disorder/sensitive skin near stimulation locations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of Depression before Transcranial direct current stimulation (tDCS) | Study tDCS Administration Visit (Day1)
  Measured by the Beck Depression Inventory (BDI-II) which is a brief, criteria-referenced assessment for measuring depression severity. The BDI-II consists of 21 items to assess the intensity of depression. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression.
Level of Anxiety before Transcranial direct current stimulation (tDCS) | Study tDCS Administration Visit (Day1)
  Measured by the Beck Anxiety Inventory (BAI) which is a brief, criteria-referenced assessment for measuring anxiety severity and level. Participants respond to 21 items rated on a scale from 0 to 3. Each item is descriptive of subjective, somatic, or panic-related symptoms of anxiety. BAI has been found to discriminate well between anxious and non-anxious diagnostic groups in a variety of clinical populations.
Intensity level of Depressive Symptoms | Study tDCS Administration Visit (Day1)
  Measured by the Hamilton Depression Rating Scale (HAM-D) which is a 17-item measure that was designed to assess frequency and intensity of depressive symptoms in patients with Major Depressive Disorder (MDD). This measure contains somatic and suicidal ideation items and has demonstrated reliability, validity, and efficiency in adult populations
Intensity level of Depressive Symptoms using SMDDS | Study tDCS Administration Visit (Day1)
  The Symptoms of Major Depressive Disorder Scale (SMDDS) is a brief self reported measure for adults with MDD and measures specific symptom dimensions. The qualitative measure has good psychometric properties including high reliability and validity.
Change in the negative affect after Transcranial direct current stimulation (tDCS) | Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
  The Positive and Negative Affect Schedule (PANAS-SF) will be administered before and after the Transcranial direct current stimulation (tDCS) session. This is a self-report questionnaire that consists of two 10-item scales (20 items total) to measure both positive and negative affect.
Change in the negative mood after Transcranial direct current stimulation (tDCS) | Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
  Will be assessed by using the Analog Mood Scale (AMS). This is a brief measure of positive and negative mood consisting of three questions (i.e., "How anxious are you?", "How sad are you?", and "How happy are you?"). Participants were told to indicate their present mood by identifying a location on a horizontal line divided into 30 equally distanced segments labeled 1 (not at all) to 30 (very much).
Change in attention bias using the Dot Probe task | Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
  The dot-probe task will be used to assess depression-related attention bias before and after tDCS administration.To complete the Dot-Probe task, participants will be shown two emotional images (e.g., sad and neutral pair or happy and neutral pair) simultaneously followed by a target in the location of one of the emotional images. Response latencies to targets replacing either the negative/positive or neutral images will be measured before and after training which will be the primary study outcome.
Change in attention bias using the Visual Search task | Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
  The Visual Search task will be administered to further assess attention bias, particularly examining the interference and facilitation effects in attention using emotional stimuli. The task uses emotional faces or words as stimuli, where the participant is instructed to search for the face that does not fit into the search set with respect to gender, where the target and distractors are expressing different or same emotions. This study will use this task as an outcome measure of Attention Bias alongside the Dot Probe task. For this task, mean response time (the time between display onset and button press) to the target stimulus for each stimulus type is measured as the main outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Kyrana Tsapkini, PhD, Principal Investigator — Johns Hopkins University